CLINICAL TRIAL: NCT05706376
Title: An Evidence-based Family Support Program for Parents and Children in Palestine: a Theory-based Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-08-7367
Record Dates: First submitted 2022-09-19; First posted 2023-01-31 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Adolescent; Psychopathology; Parent-Child Relations; Violence
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Promoting Positive Family Futures (Experimental)
  Interventions: Behavioral: Promoting Positive Family Futures
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Promoting Positive Family Futures — Promoting Positive Family Futures is a group-based program that aims to help parents and their adolescent children (13-16 yrs) cope with chronic violence by developing emotional and cognitive awareness, learning constructive conflict resolution strategies, and developing family-wide emotional security and positive family relationships. Emotional Security Theory is the foundational conceptual model for the program, and as such, the PPFF focuses on promoting family-wide communication and establishing emotional security in both the family and community across multiple sessions.Firmly grounded the cultural context of Palestine, the intervention also incorporates intervention elements derived from social ecological theories of resilience, and cognitive behavioral approaches to coping. In total, the program includes 8 sessions lasting approximately 1.5 hours each.
  Arms: Promoting Positive Family Futures
Behavioral: Treatment as Usual — Families assigned to the TAU condition will participate in a common service offered by both PCC and CRS - a weekly adolescent-only support group. Both CRS and PCC conduct extended group programs for children and adolescents (24 sessions at PCC; 25 sessions at CRS).
  Arms: Treatment as Usual

SUMMARY:
Few evidence-based programs exist to support children and families affected by sociopolitical conflict, despite documented evidence of their heightened risk for emotional and behavioral adjustment problems associated with exposure to conflict and violence at multiple levels of the social ecology (e.g., political, community, and family). Thus, a critical need exists for an evidence-based program to ameliorate the impact of political violence on the overall well-being of children and families. The current study will conduct a rigorous evaluation of a theoretically-driven, family-based intervention program in Palestine, including both the West Bank and Gaza. Firmly grounded in the cultural context of Palestine but with broad implications for individuals exposed to sociopolitical violence, the long-term goal of this project is to provide a family-focused intervention program (Promoting Positive Family Futures; PPFF) that may facilitate individuals' sense of safety and support in the context of chronic adversity. The objective is to evaluate this intervention program in the context of a randomized clinical trial (RCT) in the West Bank and Gaza (N=300). The central hypothesis is that the program will have direct positive effects on family conflict, parent psychopathology and parental security in the family as well as on adolescent emotional security in the family, with cascading effects on adolescent adjustment. Consistent with family systems theory, we further hypothesize that treatment effects on parents will mediate on the effects of the treatment on adolescent adjustment. The rationale is that bolstering resilience in family systems is a key approach to promoting positive functioning in families exposed to chronic violence. The hypothesis will be evaluated with three specific aims: 1) evaluate the efficacy of an evidence-based family support program; 2) examine process models of treatment change, and 3) examine interrelations between parent and child functioning. To achieve these aims, the study will be an RCT employing a longitudinal design (N=300) with multi-method assessments at baseline (T1), post-test (T2), 6-month follow-up (T3) and 12-month follow-up (T4). Families included in the study will be evenly divided between the West Bank (n=150) and Gaza Strip (n=150). Families will be randomized into the intervention condition (PPFF) or treatment as usual (TAU). Each territory will have an implementing partner, and implementing partners and investigators will work together to ensure the study procedures are implemented in parallel across sites. Data collection will be conducted by trained research staff from a third-party survey and policy research organization. The proposal seeks to shift current research and clinical paradigms in these contexts by employing novel theoretical concepts, approaches, and methodologies. The contribution will be significant by 1) further developing new directions for empirically-based interventions in these high-risk contexts, and 2) advancing a relatively brief, cost-effective program that can be readily implemented to help children and families exposed to continuing conflict in Palestine, with the potential to be brought to scale in other contexts.

ELIGIBILITY:
Inclusion Criteria:

* a willing adolescent between the ages of 13 and 16
* assuming a two-parent family, a mother and father willing to participate
* within the service area of implementing organizations

Exclusion Criteria:

* Families with individuals with significant mental or physical impairments precluding their ability to participate in groups

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2027-03-13 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Parental Depression | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Parental Depression will be measured using the Patient Health Questionnaire (PHQ9; Kronke & Spitzer, 2009), which has established validity in both English and Arabic, and has been successfully used in Palestinian samples (Hobfoll, et al., 2011). We hypothesize that parents in the treatment group will report lower levels of depressed mood at T2, T3 and T4 and that change in parental depression at T2 will mediate the relationship between intervention and adolescent adjustment at T3/T4.
Parental Anxiety | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Parental Anxiety will be measured using the GAD-7 (Spitzer et al., 1999), which has established validity in both English and Arabic. We hypothesize that parents in the treatment group will report lower levels of anxiety at T2, T3 and T4 and that change in parental anxiety at T2 will mediate the relationship between intervention and adolescent adjustment at T3/T4.
Parental Posttraumatic Stress | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Parent posttraumatic stress will be assessed using the PTSD Checklist - 5, which assesses symptoms of posttraumatic stress in the domains of re-experiencing, avoidance, negative mood and cognition, and hyperarousal (Weathers, et al., 2013) and has been successfully used in the region (Bensimon, Bodner, & Shrira, 2017). We hypothesize that parents in the treatment group will report lower levels of posttraumatic stress at T2, T3 and T4 that change in parental posttraumatic stress at T2 will mediate the relationship between intervention and adolescent adjustment at T3/T4.
Parent Emotional Security in Family | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Parent Emotional Security in the Family will be assessed using the Security in the Family System Scale (Forman & Davies, 2005), which has established psychometric properties and has successfully been used in other conflict settings (Cummings, et al., 2010). We hypothesize that mothers and fathers in the treatment group will report higher levels of emotional security at T2, T3, and T4 and that change parent emotional security at T2 will indirectly affect adolescent adjustment and emotional security at T3/T4.
Adolescent Security in the Family Scale | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Adolescent Emotional Security in the Family will be assessed using the Security in the Family System Scale (Forman & Davies, 2005), which has established psychometric properties and has successfully been used in other conflict settings (Cummings, et al., 2010). We hypothesize that adolescents in the treatment group will report higher levels of emotional security at T2, T3, and T4.
Adolescent Adjustment and Prosocial Skills | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Adolescent Adjustment & Prosocial Skills will be measured using the Strengths and Difficulties questionnaire, which measures children's adjustment in 5 domains: emotional symptoms, conduct problems, hyperactivity/ inattention, peer relationship problems and prosocial skills. It has been successfully validated in Arabic (Alyhari & Goodman, 2006). We hypothesize that adolescents in the treatment group will report lower levels of adjustment problems at T3/T4.
Adolescent Posttraumatic Stress Symptoms | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Adolescent Posttraumatic Stress will be assessed using the Child Posttraumatic Stress Symptom Index (Pynoos, Frederick & Nader, 1987), which has been successfully used with adolescents living in Palestine (Dubow, et al., 2012). WE hypothesize that adolescents in the PPFF condition will report lower levels of posttraumatic stress symptoms at T3 and T4.
Adolescent and Parent Resilience | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Adolescent and Parent Resilience will be assessed using the Child and Youth Resilience Measure/Adult Resilience Measure (CYRM; Ungar & Liebenberg, 2011), which assesses resilient functioning across three domains - individual resilience, relational resilience, and community resilience. The CYRM was developed in the context of a multi-national study that included a large sample drawn from Palestine, and as such, has established validity in the region (Ungar & Liebenberg, 2011). We hypothesize that adolescents in the treatment group will report higher levels of resilience at T3/T4.
Family-Wide Conflict | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Interparental and family problem solving interactions will be coded in real time for constructive and destructive conflict behaviors using the Family Interactions Coding System (FICS; Bergman and Cummings, unpublished coding system) The FICS is a well-established system for coding conflict behaviors on a 5-point scale. Inter-rater reliability for observational codes using the FICS ranges from .94 to .98. We hypothesize the the PPFF program will be associated with reductions in family-wide conflict at T2, T3, and T4 and that improvements in conflict at T2 will predict adolescent adjustment at T3/T4.
Parent-Adolescent Attachment | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Parent-Adolescent Attachment will be measured by adolescent report on the Inventory of Parent and Peer Attachment (IPPA; Greenberg & Armsden, 1987), which assesses both positive and negative dimensions of relationship quality with an attachment figure. Adolescents will complete the survey regarding their relationship with both their mother and father at all four time points of assessment. We hypothesize that adolescents in the treatment group will report improved attachment at T2, T3, and T4.
Family conflict and cohesion | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Family conflict and cohesion will be assessed using the conflict and cohesion subscales of the Family Environment Scale (Moos & Moos, 2002). All family members will complete these items at each assessment. We hypothesize that participation in the treatment condition will be associated with reduced conflict and improved cohesion for mothers, fathers, and adolescents.
Parent and adolescent emotion regulation | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Cognitive strategies for emotion regulation will be assessed using the Emotion Regulation Questionnaire (Gross & John, 2003). We hypothesize that parents and adolescents participating in PPFF will have better emotion regulation at post-test, which will in turn predict better mental health outcomes at each follow-up.
Parent and adolescent well-being | baseline, 10 week follow-up, 6 month follow-up, 12 month follow-up
  Wellbeing will be assessed using the WHO-5 Wellbeing index. We hypothesize that parents and adolescents participating in the PPFF program will have higher levels of wellbeing at all follow-up assessments as compared to the TAU group.

CONTACTS AND LOCATIONS:
Locations (1):
- University of NotreDame, Notre Dame, Indiana, United States

IPD SHARING:
Plan to Share IPD: No